CLINICAL TRIAL: NCT07312240
Title: LONgitudinal and Integrated Evaluation of Biomarkers in reLation to phenotYpe in ALS
Acronym: LONELYALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23A307
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Phenotyping; Biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Spinal Puncture; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALS Patients (Other): Patients with Amyotrophic Lateral Sclerosis
  Interventions: Diagnostic Test: Lumbar Puncture for analysis of Cerebrospinal Fluid; Diagnostic Test: Deep Phenotyping; Diagnostic Test: Routine blood chemistry analysis and genetic analysis
- Controls (Other): Individuals undergoing Lumbar Puncture for neurological symptoms but finally having no evidence of nervous system pathology
  Interventions: Diagnostic Test: Lumbar Puncture for analysis of Cerebrospinal Fluid

INTERVENTIONS:
Diagnostic Test: Lumbar Puncture for analysis of Cerebrospinal Fluid — Lumbar Puncture for analysis of Cerebrospinal Fluid for subsequent discovery and validation of a novel biomarker
Diagnostic Test: Deep Phenotyping — Clinical, neurophysiological, neuroradiological, neuropsychological phenotyping and respiratory investigation
  Arms: ALS Patients
Diagnostic Test: Routine blood chemistry analysis and genetic analysis — Plasma sampling and genetic analysis
  Arms: ALS Patients

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease characterized by progressive degeneration of upper and lower motor neurons, leading to paralysis and death. Despite its uniformly fatal outcome, ALS shows marked clinical heterogeneity with respect to phenotype, progression rate, cognitive involvement, and survival. This heterogeneity limits prognostic accuracy and complicates patient stratification in both clinical practice and research settings.

Neurochemical biomarkers have emerged as promising tools to improve diagnosis, prognostication, and understanding of ALS pathophysiology. Among them, neurofilament light chain (NfL) represents the most established biomarker, reflecting axonal degeneration. Additional biomarkers, including glial fibrillary acidic protein (GFAP), phosphorylated tau (p-tau181), and Alzheimer's disease-related markers (Aβ42 and Aβ40), may provide complementary information regarding astroglial activation, motor neuron subtype involvement, and cognitive-behavioral features. However, the phenotypic correlates, longitudinal trajectories, and biological determinants of these biomarkers in ALS are not yet fully understood.

The LONELYALS study is an ongoing, monocentric, observational cohort study with a case-control component, designed to investigate the relationships between ALS phenotype and a comprehensive panel of cerebrospinal fluid (CSF) and blood biomarkers. The study will enroll 140 adult patients with ALS and collect longitudinal clinical, neuropsychological, biological, and laboratory data over a follow-up period of up to 36 months. By integrating biomarker measurements with detailed phenotypic characterization, the study aims to clarify biomarker origins, determinants, and prognostic value, and to identify novel CSF biomarkers relevant to ALS.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disorder affecting upper and lower motor neurons and leading to muscle weakness, paralysis, and premature death. Although ALS is uniformly fatal, it is characterized by substantial clinical and biological heterogeneity, including differences in site of onset, rate of disease progression, cognitive and behavioral involvement, and survival. This heterogeneity poses major challenges for prognostication, patient counseling, and the design and interpretation of clinical trials.

In recent years, neurochemical biomarkers have gained increasing relevance in ALS research. Neurofilaments, particularly neurofilament light chain (NfL), are currently the most widely studied biomarkers and are considered indicators of axonal degeneration. Elevated NfL levels in cerebrospinal fluid (CSF) and blood have been consistently observed in ALS and are associated with disease severity and survival. However, several key questions remain unresolved, including the relative contribution of upper versus lower motor neuron degeneration to NfL release, the extent to which NfL reflects disease aggressiveness versus anatomical disease burden, and the factors influencing its distribution between CSF and blood.

Other biomarkers may capture complementary aspects of ALS pathophysiology. Glial fibrillary acidic protein (GFAP), a marker of astrocytic activation, has been reported to be increased in ALS and may be related to extra-motor and cognitive features. Phosphorylated tau (p-tau181), widely used as a biomarker of Alzheimer's disease, has recently been proposed as a potential ALS biomarker, possibly reflecting lower motor neuron degeneration. In addition, classic Alzheimer's disease biomarkers such as Aβ42 and Aβ40 may provide insights into cognitive impairment and overlapping neurodegenerative mechanisms in ALS. The relationships among these biomarkers, their longitudinal evolution, and their associations with clinical phenotype and disease progression remain insufficiently characterized.

The LONELYALS study (LONgitudinal and integrated Evaluation of biomarkers in reLation to phenotYpe in ALS) is an ongoing, monocentric, observational clinical-epidemiological study focusing on biological material. The study adopts a prospective cohort design with a case-control component and is conducted at a single specialized ALS center. A total of 140 adult patients with ALS, aged 18 to 90 years, are being enrolled and followed longitudinally for up to 36 months. Patients are recruited during inpatient admissions, and all participants provide biological samples and clinical data according to standardized procedures.

The study involves the collection and analysis of CSF and blood samples, including genetic material, alongside comprehensive clinical, neurological, and neuropsychological assessments. Biomarkers of interest include established and emerging neurochemical markers related to axonal degeneration, astroglial activation, tau pathology, and amyloid metabolism. Longitudinal sampling allows evaluation of biomarker trajectories over time and their relationship with disease progression.

The primary objectives of the study are to explore the associations between baseline biomarker levels and ALS phenotype, to assess the relationships between CSF and blood biomarker concentrations, and to evaluate the prognostic value of biomarkers with respect to longitudinal clinical evolution. Additional aims include investigating the influence of physiological and pathophysiological factors-such as age, sex, body mass index, and renal function-on biomarker levels; exploring interrelationships among different biomarkers; and identifying novel CSF biomarkers relevant to ALS.

By integrating longitudinal biomarker data with detailed phenotypic characterization, the LONELYALS study seeks to improve understanding of ALS pathophysiology and heterogeneity. The results are expected to support biomarker-based patient stratification, facilitate more accurate prognostication, and contribute to the development of personalized clinical management strategies. In the longer term, improved biomarker characterization may also enhance patient selection and outcome assessment in future interventional trials.

ELIGIBILITY:
Inclusion Criteria ALS patients:

* diagnosis of Amyotrophic Lateral Sclerosis (ALS);
* age ≥18 y;
* feasibility of lumbar puncture (LP);
* informed consent.

Exclusion Criteria ALS patients:

* severe medical comorbidities;
* recent traumatic, inflammatory, vascular, or neoplastic Central Nervous System disease; contraindications to LP.

Inclusion Criteria Controls:

* age ≥18 y;
* individuals undergoing LP for neurological symptoms;
* no evidence of nervous system pathology;
* informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Clinical - ALSFRS-R score | At enrolment, at 6 months, at 12 months
Clinical - Penn UMN Score | At enrolment, at 6 months, at 12 months
Clinical - LMN score | At enrolment, at 6 months, at 12 months
Neuropsychological phenotyping | At enrollment
  Score at Montreal Cognitive Assessment
Neurophysiological - Limb denervation score (EMG) | At enrollment
Neurophysiological - CMCT (central motor conduction time) (TMS, transcranial magnetic stimulation) | At enrolment
Arterial blood gas analysis - PaO2 | At enrollment
Arterial blood gas analysis - PaCO2 | At enrolment
Neuroradiological phenotyping | At enrollment
  Presence or absence of T2-FLAIR hyperintensity of the corticospinal tracts
Neurochemical - Plasma NFL | An enrolment, at 6 months, at 12 months
Outcome measure for controls | At enrolment
  Exclusion of ALS or other neurodegenerative diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy